CLINICAL TRIAL: NCT02981316
Title: Treatment of Recurrent Clostridium Difficile Infection With RBX7455: A Dose-ranging, Prospective, Single Center, Open Label Phase I Trial
Brief Title: Treatment of Recurrent Clostridium Difficile Infection With RBX7455
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Rebiotix Inc. (Industry)
Responsible Party: Principal Investigator, Sahil Khanna, M.B.B.S., Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-008828
Record Dates: First submitted 2016-12-01; First posted 2016-12-05 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Clostridium Difficile Infection
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- RBX7455 Group A (Active Comparator): 4 days of 4 capsules twice daily RBX7455 for 10 subjects.
  Interventions: Biological: RBX7455
- RBX7455 Group B (Active Comparator): 2 days of 4 capsules twice daily RBX7455 for 10 subjects.
  Interventions: Biological: RBX7455
- RBX7455 Group C (Active Comparator): 2 days of 2 capsules twice daily RBX7455 for 10 subjects.
  Interventions: Biological: RBX7455
- RBX7455 Group D (Active Comparator): 2 days of 1 capsule twice daily RBX7455 for 10 subjects.
  Interventions: Biological: RBX7455

INTERVENTIONS:
Biological: RBX7455 — Microbiota capsule(s) given twice daily in the morning, and in the evening.

SUMMARY:
The purpose of this study is to demonstrate the efficacy and safety of RBX7455 for the treatment of recurrent CDI in subjects who have had at least one recurrence after a primary episode (i.e., at least two episodes) and have completed at least two rounds of standard-of-care oral antibiotic therapy.

ELIGIBILITY:
Inclusion criteria:

1. ≥ 18 years old.
2. Medical record documentation of recurrent CDI, defined as at least one recurrence after a primary episode and has completed at least two rounds of standard-of-care oral antibiotic therapy. Study subjects will have their diarrhea resolved, i.e., would be having less than 3 watery bowel movements at the time of study enrollment for 48 hours or more.
3. A positive stool test for the presence of C. difficile within 30 days prior to enrollment and standard C. difficile treatment.
4. Willing and able to swallow capsules.
5. Agrees to abstain from non-dietary probiotics for the duration of the study.
6. Agrees to abstain from vancomycin, metronidazole, fidaxomicin, rifaximin, nitazoxanide and IVIG for the duration of the study unless prescribed to treat recurrent CDI.
7. Agrees to stop proton pump inhibitors or H2 blocker medications.
8. Agrees to practice a form of effective contraception during study participation.
9. Has a negative urine pregnancy test at the time of enrollment (females of child-bearing potential only).
10. Willing and able to provide informed consent and HIPAA authorization.
11. Willing and able to complete the required Subject Diary.
12. Willing and able to meet all study requirements, including attending all assessment visits and phone calls.

Exclusion criteria:

1. A known history of continued CDI diarrhea, despite being on a course of antibiotics prescribed for CDI treatment.
2. Requires continuous antibiotic therapy for a condition other than CDI.
3. Previous fecal transplant.
4. Previous treatment with RBX2660.
5. Diagnosis of inflammatory bowel disease (IBD), e.g., ulcerative colitis, Crohn's disease, or microscopic colitis.
6. Diagnosis of irritable bowel syndrome (IBS) as determined by Rome III criteria.
7. History of chronic diarrhea.
8. History of celiac disease.
9. Disease symptoms caused by a confirmed intestinal pathogen other than C. difficile.
10. Unable to stop proton pump inhibitors or H2 blocker medications.
11. Colostomy.
12. Intra-abdominal surgery within the last 60 days.
13. Evidence of active, severe colitis.
14. History of short gut syndrome.
15. Requires the regular use of medications to manage bowel hypermotility.
16. Planned therapy in the next 3 months that may cause diarrhea (e.g., chemotherapy).
17. Planned surgery requiring perioperative antibiotics within 3 months of study enrollment.
18. Life expectancy of < 6 months.
19. Compromised immune system (e.g., HIV infection; AIDS-defining diagnosis or CD4 <200/mm3; inherited/primary immune disorders; immunodeficient or immunosuppressed due to a medical condition or medication; current or recent (< 90 days) treatment with chemotherapy; or current or recent (< 90 days) treatment with immunosuppressant medications.
20. Taking systemic steroids (≥ 20 mg a day or prednisone-equivalent) or is expected to be on steroids after enrollment through 8 weeks after completing the assigned study treatment.
21. An absolute neutrophil count of <1000 cells/µL.
22. Known or suspected current (< 90 days) illicit drug use. Note: marijuana use is allowed.
23. Pregnant, breastfeeding, or intends to become pregnant during study participation.
24. Participating in a clinical trial of another investigational product (drug, device or other) and has not completed the required follow-up period.
25. Subject, in the opinion of the investigator, for whatever reason, should be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-11; Primary Completion 2020-07-22 (Actual); Study Completion 2020-07-22 (Actual)

PRIMARY OUTCOMES:
Time to recurrence of Clostridium Difficile Infection (CDI) | approximately 8 weeks
Number of patients experiencing adverse events | approximately 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sahil Khanna, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khanna S, Pardi DS, Jones C, Shannon WD, Gonzalez C, Blount K. RBX7455, a Non-frozen, Orally Administered Investigational Live Biotherapeutic, Is Safe, Effective, and Shifts Patients' Microbiomes in a Phase 1 Study for Recurrent Clostridioides difficile Infections. Clin Infect Dis. 2021 Oct 5;73(7):e1613-e1620. doi: 10.1093/cid/ciaa1430. PMID 32966574
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials